CLINICAL TRIAL: NCT07072741
Title: Assessing the Feasibility and Acceptability of Watching Queen of Katwe as a Role Model Intervention Among Adolescents in High Schools in Kenya
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shamiri Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Shamiri Queen of Katwe Project
Record Dates: First submitted 2025-06-30; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Observational Study
Keywords: Queen of Katwe; Media-based intervention; Role model intervention; Film-based learning; Low-cost intervention; Adolescent motivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shamiri Queen of Katwe (Experimental): The session itself will take approximately two hours-this includes student assembly, an introduction to the study, and the screening of Queen of Katwe
  Interventions: Other: Shamiri Queen of Katwe Intervention

INTERVENTIONS:
Other: Shamiri Queen of Katwe Intervention — The intervention involves screening the film Queen of Katwe to high school students in a school setting.

SUMMARY:
This study will test whether using the film Queen of Katwe as a role model story can help motivate and engage high school students in Kenya. The film is based on the true story of Phiona Mutesi, a Ugandan girl who becomes a chess champion despite growing up in poverty. The study will take place in a mixed secondary school in Ngong town, Kajiado County, with about 250 students aged 13 to 19. Students will watch the film at school. To see if the approach works well, researchers will collect data before and after the film showing.

They will check:

1. Feasibility (how easy it is to carry out, including costs and logistics)
2. Acceptability (how students and teachers feel about it)
3. Engagement (how involved students are) Surveys and focus groups will be used to gather feedback. The goal is to see if this low-cost method could be used more widely to support learning and motivation in schools.

DETAILED DESCRIPTION:
This study examines the feasibility and acceptability of using the film Queen of Katwe-which tells the true story of Phiona Mutesi, a Ugandan girl from an underprivileged background who becomes a chess champion-as a role model intervention to inspire motivation and academic engagement among adolescents in high school students in Kenya. Media-based interventions have gained recognition as effective tools for promoting student learning and well-being, yet their implementation in school settings remains underexplored. This study will employ a feasibility study design and be conducted in a mixed secondary school in Ngong town, Kajiado County, Kenya, with a sample of ~250 students aged 13-19 years. Students will watch Queen of Katwe in their school setting, and data will be collected before and after the intervention to assess feasibility, acceptability, and engagement. Feasibility will be evaluated based on logistical observations, cost analysis, and the Feasibility of Intervention Measure. Acceptability will be assessed through a screening survey using the Acceptability of Intervention Measure, while focus group discussions with students and teachers will provide qualitative insights. The findings will offer valuable evidence on the potential of media-based interventions to enhance motivation and academic engagement in Kenyan schools. If found feasible and acceptable, this low-cost, scalable approach could inform future educational policies and programs aimed at supporting student aspirations and learning outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be high school students in the selected school.
* Participants must be between the ages of 13 to 19.

Exclusion Criteria:

* There will be no other exclusion criteria.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-07-23 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in aspiration score from baseline on the Aspirations Index through study completion | From baseline through endline, an average of two days
  Changes in self-reported aspirations as measured by the Aspiration Index is used to assess long term aspirations and goals that individuals hope to accomplish in their lives. In this study, we will use a shortened 15-item version of this scale including items on aspirations of wealth, fame, image, personal growth, relationship, community and health. The scores for each item ranges between 1-7, with higher scores indicating higher aspirations.
Mean change in school engagement score from baseline on the School Engagement Measure through study completion. | From baseline through endline, an average of two days
  Changes in self-reported school engagement as measured by the School Engagement Measure refer to a student's emotional, behavioural, and cognitive involvement in school activities and learning. This is a 19-item measure with responses measured on a 5-point Likert scale ranging from 1 (not at all true) to 5 (very true). Higher scores indicate greater school engagement.
Change in academic performance as measured using the average grades | Periprocedural - From academic exam results pre-intervention to academic exam results post-intervention, up to three months
  Changes in academic performance as measured using the average grades obtained from the most recent exam prior to the intervention, and the first available exam following the implementation of the intervention.
Mean score of the Feasibility of Intervention Measure at study completion | At study completion, up to three months
  Feasibility of Intervention Measure tracks metrics such as ease of setting up the screenings, logistical challenges, and time constraints. It assesses the extent to which an intervention can be successfully implemented within a given setting. This is a 4-item measure with responses measured on a 4-point Likert scale ranging from 1 (Completely disagree) to 5 (Completely agree). Higher scores indicate a better outcome, good scores on the feasibility of the intervention.
Mean score of the Acceptability of Intervention Measure at study completion | At study completion, up to three months
  Acceptability of Intervention Measure assess the acceptability of the intervention by participants. This 4-item measure evaluates stakeholders' perception of an intervention's acceptability, determining whether they find it agreeable, satisfactory, or palatable. Responses are measured on a 4-point Likert scale ranging from 1 (Completely disagree) to 5 (Completely agree). Higher scores indicate a better outcome, the acceptability of the intervention.
Mean score of the Intervention Appropriateness Measure at study completion | At study completion, up to three months
  Intervention Appropriateness Measure assesses perceptions of participants' intervention appropriateness. It measures the perceived fit, relevance, or compatibility of an intervention within a particular context. This 4-item measure determines whether an intervention aligns with the needs of a specific population, organisational goals, or existing workflows. Responses are measured on a 4-point Likert scale ranging from 1 (Completely disagree) to 5 (Completely agree). Higher scores indicate a better outcome, the appropriateness of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tom L Osborn, Principal Investigator — Shamiri Institute
Locations (1):
- Shamiri Institute, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
The investigators intend to share fully de-identified data through publications and upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 3 years following article publication.
Access Criteria: Access to study reports and protocols will be open. Access to de-identified individual participant data will be available upon request from the study team.